CLINICAL TRIAL: NCT01801306
Title: A New Multi-parameter Monitoring System Applying Near Infrared Spectroscopy and Indocyanine Green to Detect Cerebrovascular Events in Patients With Subarachnoid Hemorrhage
Brief Title: A New Minimal-invasive Brain Tissue Probe Applying Near Infrared Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeMoDevices AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIV-12-04-006261
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NeMoProbe (Other): The NeMo System is used for intracranial pressure (ICP) and brain temperature monitoring, as well as the determination of the brain tissue oxygenation saturation (SbtO2) and cerebral blood flow. The sensors for NIRS are implemented into a conventional brain tissue probe for ICP monitoring (NeMo Probe).
  Interventions: Device: NeMo Probe

INTERVENTIONS:
Device: NeMo Probe — A new minimal-invasive brain tissue probe applying near infrared spectroscopy

SUMMARY:
To assess the feasibility of a new brain tissue probe for multi-parameter neuromonitoring (NeMo Probe) and the accuracy of measurement values.

To demonstrate the ability of the NeMo probe to detect changes in cerebral hemodynamics and oxygenation during cerebrovascular events monitored with established methods including brain tissue oxygenation tension and microdialysis

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-75 years (inclusive)
* Patients with high-grade subarachnoid hemorrhage (WFNS 4-5)
* Decreased level of consciousness with the need for intracranial pressure monitoring
* Successful exclusion of the ruptured aneurysm with clipping or coiling
* Women of childbearing potential must have a negative serum pregnancy test
* Written informed consent obtained by a legal representative

Exclusion Criteria:

* Significant kidney and/or liver disease
* Any severe unstable concomitant condition or disease (e.g. cancer, coronary disease) or chronic condition (e.g. psychiatric disorder, chronic obstructive pulmonary disease Grade II, chronic heart failure > NYHA II)
* Cerebrospinal fluid infection or signs of meningoencephalitis
* Acute respiratory distress syndrome (ARDS), pulmonary edema
* Preexisting coagulation disorder
* Patients with current alcohol or drug abusus or dependence
* Patients with a history of hypersensitivity against indocyanine green or sodium iodine
* Patients with thyroid disease causing hyperthyroidism
* Breast-feeding women
* Patients committed to an institution based on official directive or court order

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To assess the feasibility of the neuromonitoring system and accuracy of the measurement values | Day 90 after Removal of Medical Device
  Feasibility: User acceptance rate in comparison to conventional probes for ICP-monitoring. The following parameters will be analysed:
  * Incidence of concerns of users in relation to the installation of the NeMo System
  * Incidence of concerns of users in relation to the function of the NeMo System Incidence of concerns of users in relation to the removal of the NeMo System
  * User-friendliness with a 3-graded scale (equal, better, worse) compared to conventional probes for ICP monitoring Accuracy of measurement values: Results from repeated measurements of mttICG, CBV, and CBF.
  Safety endpoints:
  -Adverse events profile (including adverse device effects): Incidence of complications (infections, brain tissue damage, hemorrhage) in comparison to historical series (conventional probes for ICP-monitoring):

SECONDARY OUTCOMES:
To demonstrate the ability of the neuromonitoring system to detect cerebrovascular events in patients with subarachnoid hemorrhage | Day 90 after Removal of Medical Device
  Results concerning the response to cortical spreading depolarization (CSD) monitored with electrocorticography (ECoG):
  Increase of brain tissue oxygenation (SbtO2), total hemoglobin (dHbtotal, aHbtotal), CBV, CBV Hb and CBF >20% Decrease of SbtO2, dHbtotal, aHbtotal, CBV, CBV Hb and CBF >20% Changes of SbtO2, dHbtotal, aHbtotal, CBV, CBV Hb and CBF <20%
  Results concerning the sensitivity and specificity to detect delayed cerebral ischemia (DCI) monitored with ptiO2 and MD:
  Correlation of CBF values <15 ml/100g/min with defined criteria for DCI (ptiO2 <15 mmHg, Gluc brain<0.7 mmol/l, Lactate-Pyruvate-Ratio >40), number of false negative and false positive events, Receiver Operating Characteristic (ROC) curve.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Seule, MD, Principal Investigator — Department of Neurosurgery, University Hospital Heidelberg
Locations (1):
- Department of Neurosurgery, University Hospital Heidelberg, Heidelberg, Germany